CLINICAL TRIAL: NCT03084315
Title: Changes in Biomarkers Associated With Use of Electronic Cigarettes Among African American Menthol and Nonmenthol Smokers
Brief Title: Changes in Biomarkers Associated With Use of Electronic Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2015NTLS139
Record Dates: First submitted 2017-03-13; First posted 2017-03-20 (Actual); Results first posted 2020-03-20 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Biomarkers
Keywords: smoking; electronic cigarettes; nicotine
MeSH Terms: conditions — Smoking; Vaping | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Intervention Model Description: Blocked randomization, block size unknown to staff or investigators
Who Masked: Participant
Masking Description: All participants are blinded to intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- E-Cig Zero Nicotine (Sham Comparator): E-Cigarette with no nicotine added
  Interventions: Device: E-Cig Zero Nicotine
- E-Cig 24mg Nicotine (Active Comparator): E-cigarette with 24mg of nicotine added
  Interventions: Device: E-Cig 24mg Nicotine

INTERVENTIONS:
Device: E-Cig Zero Nicotine — E-Cig Zero Nicotine
  Arms: E-Cig Zero Nicotine
Device: E-Cig 24mg Nicotine — E-Cig 24mg Nicotine
  Arms: E-Cig 24mg Nicotine

SUMMARY:
The objective of this clinical trial was to compare the effects of e-cigarettes with and without nicotine on patterns of combustible cigarette use and biomarkers of exposure to tobacco toxicants among African American smokers.

DETAILED DESCRIPTION:
This study compares patterns of e-cigarette use and the exposure to the tobacco-specific carcinogen 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) in African American smokers, randomized to ad lib e-cigarettes containing nicotine vs. no nicotine. We hypothesized that nicotine e-cigarettes would be used more than no-nicotine e-cigarettes, and that this would be associated with reduced use of combustible cigarettes. We hypothesized that nicotine e-cigarettes would result in more substitution for combusted cigarettes than no-nicotine e-cigarettes and result in lower levels of exposure to the tobacco-specific carcinogen NNAL. These results would be relevant for developing exposure reduction strategies for adult African American smokers.

ELIGIBILITY:
Inclusion Criteria:

1. self-identify as African American or Black;
2. age 18 years or older;
3. smoke at least five cigarettes daily for the past year;
4. not interested in quitting smoking in the next 6 months;
5. Willing to use e-cigarettes;
6. Good physical health (no unstable medical or mental health condition);
7. no contraindications for e-cigarette use.

Exclusion Criteria:

1. Recent unstable or untreated psychiatric diagnosis including substance abuse, as determined by the DSM-IV criteria;
2. use in the past 30 days of tobacco or nicotine products including e-cigarettes, other than regular cigarettes;
3. participation in a smoking cessation program in the past 30 days;
4. pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Joseph, MD, Principal Investigator — University of Minnesota
Locations (1):
- DCRU, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Okuyemi KS, Ojo-Fati O, Aremu TO, Friedrichsen SC, Grude L, Oyenuga M, Shyne M, Murphy SE, Hatsukami D, Joseph AM. A Randomized Trial of Nicotine versus No-nicotine E-cigarettes Among African American Smokers: Changes in Smoking and Tobacco Biomarkers. Nicotine Tob Res. 2022 Mar 1;24(4):555-563. doi: 10.1093/ntr/ntab212. PMID 34669956

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | E-Cig Zero Nicotine | E-Cig 24mg Nicotine
Started | 116 | 118
Completed | 106 | 109
Not Completed | 10 | 9
Not completed — Lost to Follow-up | 8 | 7
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Population: 2 participants in each group withdrew from the study and were not included in the baseline characteristic data.
Groups:
- Total: Total of all reporting groups
Arm/Group | E-Cig Zero Nicotine | E-Cig 24mg Nicotine | Total
Number analyzed (Participants) | 114 | 116 | 230
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 107 | 112 | 219
  >=65 years | 7 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.74 (11.65) | 50.89 (10.74) | 50.81 (11.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 51 | 101
  Male | 64 | 65 | 129
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 111 | 113 | 224
  White | 0 | 0 | 0
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 114 | 116 | 230

OUTCOME MEASURES:

1. Primary Outcome: Change in Biomarker Concentrations: Nicotine Equivalents
Description: Change in concentration of nicotine equivalents in units of mmol/mg creatinine.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: mmol/mg creatinine
Arm/Group | E-Cig Zero Nicotine | E-Cig 24mg Nicotine
Number analyzed (Participants) | 114 | 116
mmol/mg creatinine | 74.9 (57.23) | 79.56 (72.8)

2. Primary Outcome: Change in Biomarker Concentrations: NNAL
Description: Change in urinary concentration of 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) in units of pmol/mg creatinine.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: pmol/mg creatinine
Arm/Group | E-Cig Zero Nicotine | E-Cig 24mg Nicotine
Number analyzed (Participants) | 106 | 109
pmol/mg creatinine | 1.98 (1.74) | 1.95 (1.47)

3. Other Pre Specified Outcome: Change in Average Cigarettes Per Day
Description: Participants will record the average number of cigarettes smoked per day in the 7 days leading up to each study visit. Outcome is reported as the change in average cigarettes per day from baseline to 6 weeks of treatment.
Time Frame: Baseline, Week 6
Measure: Mean (Standard Deviation); unit: cigarettes/day
Arm/Group | E-Cig Zero Nicotine | E-Cig 24mg Nicotine
Number analyzed (Participants) | 114 | 116
cigarettes/day | 8.8 (6.3) | 8.6 (6.3)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | E-Cig Zero Nicotine | E-Cig 24mg Nicotine
All-Cause Mortality (participants affected / at risk) | 0/106 | 0/109
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/109
Other Adverse Events (participants affected / at risk) | 0/106 | 0/109

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/15/NCT03084315/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT03084315/ICF_001.pdf